CLINICAL TRIAL: NCT03777085
Title: Multicenter, Randomized, Double-blind, Parallel Controlled, Phase III Clinical Study to Compare the Efficacy and Safety of TQB2303 in Conbination With CHOP Regimen (T-CHOP) Versus Rituximab in Combination With CHOP Regimen (R-CHOP) in Previously Untreated Subjects With CD20-Positive Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: Study of TQB2303 in Patients With CD20-Positive Diffuse Large B-cell Lymphoma (DLBCL)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TQB2303-III-01
Record Dates: First submitted 2018-12-13; First posted 2018-12-17 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2303 (Experimental)
  Interventions: Drug: TQB2303
- Rituximab (Active Comparator)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: TQB2303 — 375mg/m2, iv q3w,6 cycles(each cycle is 3 weeks
  Arms: TQB2303
Drug: Rituximab — 375mg/m2, iv q3w,6 cycles(each cycle is 3 weeks
  Arms: Rituximab

SUMMARY:
The Purpose of This Study is to Compare the Efficacy, Safety, Immunogenicity and Pharmacokinetics between TQB2303 and Rituximab in Combination With CHOP in Previously Untreated Patients with Diffuse Large B-cell Lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. Untreated CD20-positive DLBCL patients confirmed by histopathology or cytology.
2. 18 years to 75 years; Male or female patients.
3. International Prognostic Index (IPI) score of 0 to 2.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
5. More than 6 months life expectancy judged by the researchers.
6. At least one measurable lesions: for nodal tumor mass, more than 1.5 cm in the long axis and more than 1.0 cm in the short axis; for extranodal tumor mass, more than 1.0 cm in the long axis.
7. left ventricular ejection fraction (LVEF) measured by the Cardiac echocardiography greater than or equal to 50%.
8. Adequate hematologic function, no matter the bone marrow was attacked or not, as follows:absolute neutrophil count (ANC) ≥1.5×10^9/L and platelet count≥75×^9/L.
9. Understood and Signed an informed consent form.

Exclusion Criteria:

1. Known allergic reactions against human or murine monoclonal antibody, murine products, or foreign proteins.
2. Known allergic reactions against any component of CHOP regimen.
3. Previous treatment for DLBCL, including chemotherapy, immunotherapy, partial radiotherapy for lymphoma, or surgical treatment (excluding tumor mass biopsies and surgical resection for non-lymphoma lesions), or prior use of any monoclonal antibody within 3 month.
4. T-cell/histiocyte-rich large B-cell lymphoma, Primary DLBCL of the CNS, Primary cutaneous DLBCL, leg type, EBV-positive DLBCL of the elderly (EBV + DLBCL), EBV-positive DLBCL of the elderly (EBV + DLBCL), DLBCL associated with chronic infammation, Lymphomatoid granulomatosis, Primary mediastinal (thymic) large B-cell lymphoma (PMBL), ALK-positive large B-cell lymphoma, ALK-positive large B-cell lymphoma, ALK-positive large B-cell lymphoma, high-grade B-cell lymphoma (high-grade B-cell lymphoma with MYC, with or without concurrent in BCL2 and/or BCL6 gene rearrangements, high-grade B-cell lymphoma, NOS), B-cell lymphoma, Not categorizable, Characteristics between DLBCL and classical Hodgkin's lymphoma, transformed DLBCL, DLBCL secondary central nervous system invasion;
5. Other malignant tumors that have been or are currently suffering (healed skin basal cell carcinoma or cutaneous squamous cell carcinoma, or cutaneous melanoma or cervical carcinoma in situ).
6. Significantly poorly controlled diseases that can affect adherence to the study protocol, such as severe cardiovascular disease (such as the New York Heart Association class III or IV heart disease, myocardial infarction or unstable arrhythmia in the last 6 months or Unstable angina, severe hypertension, peripheral nervous system or central nervous system disease;
7. Patients with a history of progressive multifocal leukoencephalopathy.
8. Continuous corticosteroid treatment being received, dose >30 mg/day prednisone or equivalent dose of corticosteroids ≥10 days.
9. Participation in another interventional clinical trial in the past 3 months.
10. Patients who received or underwent major surgeries within 28 days prior to enrollment, or patients with unsurgical wounds.
11. Treated with transfusion, erythropoietin (EPO), granulocyte colony-stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF) within 14 days prior to enrollment.
12. Vaccination within 28 days or planned prior to enrollment.
13. Appearing the following laboratory abnormal values.

    1. Coagulation function: partial prothrombin time (PTT) or activated partial thromboplastin time (aPTT) or international normalized ratio (INR) > 1.5 times ULN without anticoagulant therapy.
    2. Liver function: total bilirubin (TBIL) > 1.5 times the upper limit of normal (3 times the upper limit of normal value when the liver is invaded), alanine aminotransferase (ALT) and / or aspartate aminotransferase (AST) > 2.5 times the upper limit of normal value (>5 times the upper limit of normal value when the liver is invaded)
    3. Renal function: serum creatinine (Cr) > 1.5 times the upper limit of normal value.
14. an active infection at the time of enrollment, or any major infection events that affected the enrollment of the subjects determined by the investigator within 28 days (except for neoplastic fever).
15. Suspected active or latent tuberculosis infections.
16. HBsAg positive and/or HBcAb positive and HBV DNA positive.
17. HCV antibody and HCV-RNA positive; or HIV positive patients.
18. Pregnancy or breast feeding. Companion for women of childbearing age or women of childbearing age,who reluctant to take appropriate contraceptive methods within one year after the last treatment of the study;Pregnancy before pregnancy screening, the women who blood / urine results were positive.
19. Patients that researchers deem as not appropriate to enter the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2019-01-10 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 18 weeks

SECONDARY OUTCOMES:
Objective Response Rate (CR+CRu) | 18 weeks
Progression-free survival (PFS) | 18 weeks
Event-free survival (EFS) | 18 weeks
Duration of Response (DOR) | 18 weeks
:Overall survival (OS) | 18 weeks

CONTACTS AND LOCATIONS:
Locations (31):
- China (31):
  - No.150 Haping Road, Nangang District, Haerbin, Heilongjiang
  - No. 42 Baiziting Road, Xuanwu District, Nanjing, Jiangsu
  - No.8 Jiangtan Road,Weibin District, Baoji
  - No. 87 Xiangya Road Furong District, Changsha
  - No.138 Tongzipo Road Yuelu District, Changsha
  - No.139 Renmin Middle Road Furong District, Changsha
  - No. 37 Guoxue Lane Wuhou District, Chengdu
  - No. 55 Section 4 Renmin South Road Wuhou District, Chengdu
  - No. 10 Daping Yangtze River Branch Road Yuzhong District, Chongqing
  - No.183 Xinqiao Main Street Shapingba District, Chongqing
  - No.420 Fuma Road, Jin'an district, Fuzhou
  - No.295 Xichang Road, Wuhua District, Kunming
  - No. 701 Donggang Road (West) Chengguan District, Lanzhou
  - No. 82 Cuiyingmen Chengguan District, Lanzhou
  - No.333 Nanbinhe Middle Road Qilihe District, Lanzhou
  - No. 8 Wenchang Road Chengzhong District, Liuchow
  - No.519 Beijing East Road High - tech District, Nanchang
  - No.71 Embankment Road, Qingxiu District, Nanning
  - No.20 Xisi Road Chongchuan District, Nantong
  - No.1677 Wutai Mountain Road Huangdao District, Qingdao
  - No 137 Carp mountain Road New district, Ürümqi
  - No. 151 Guangwen Street Kuiwen District, Weifang
  - No. 3, West Mt. East Road, Wendeng District, Weihai City, Weihai
  - No. 1277 Jiefang Avenue Jianghan District, Wuhan
  - No.31 Hygienic Lane Haizang Road Liangzhou District, Wuwei
  - No. 15 West ChangLe Road New City District, Xi'an
  - No.256 Youyi West Road Beilin District, Xi'an
  - No. 7 Weiwu Road Jinshui District, Zhengzhou
  - No.1 Jianshe East Road Erqi District, Zhengzhou
  - No.127 Dongming Road, Jinshuii District, Zhengzhou
  - No. 54 Communist Youth League Road Zhangdian District, Zibo